CLINICAL TRIAL: NCT04032366
Title: Inhaled Nitric Oxide as Salvage Treatment of Hypoxemia After Type A Acute Aortic Dissection Surgery (INSTEAD)
Brief Title: iNO as Salvage Treatment of Hypoxemia After TAAD Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: INSTEAD
Record Dates: First submitted 2019-07-16; First posted 2019-07-25 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-07

CONDITIONS: Type A Aortic Dissection
Keywords: Hypoxemia; Type A acute aortic dissection; inhaled nitric oxide
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood and serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PEEP 5: post-surgical type A acute aortic dissection patients was ventilated with a PEEP of 5cm H2O, without inhaled nitric oxide
- PEEP 10: post-surgical type A acute aortic dissection patients was ventilated with a PEEP of 10cm H2O, without inhaled nitric oxide
  Interventions: Drug: inhaled nitric oxide; Device: PEEP
- PEEP 10 +iNO: post-surgical type A acute aortic dissection patients was ventilated with a PEEP of 10cm H2O, with inhaled nitric oxide
- PEEP 5 +iNO: post-surgical type A acute aortic dissection patients was ventilated with a PEEP of 5cm H2O, with inhaled nitric oxide
  Interventions: Drug: inhaled nitric oxide; Device: PEEP

INTERVENTIONS:
Drug: inhaled nitric oxide — using of inhaled nitric oxide
  Other Names: iNO
  Groups: PEEP 10; PEEP 5 +iNO
Device: PEEP — increasing PEEP or decreasing PEEP
  Groups: PEEP 10; PEEP 5 +iNO

SUMMARY:
The purpose of this study was to clarify the possible mechanism of hypoxemia after surgical treatment of type A acute aortic dissection and the possible mechanism of the treatment role of inhaled nitric oxide in refractory hypoxemia.

DETAILED DESCRIPTION:
The investigators' previous study has stressed that inhaled nitric oxide therapy might play an ameliorative role in patients with refractory hypoxemia after surgical treatment of type A acute aortic dissection. The possible reason might be the decreasing of intrapulmonary shunt because previous studies showed that inhaled nitric oxide could decrease intrapulmonary shunt by selectively dilating the pulmonary vessels in ventilated areas. As a result, the investigators designed this observational study to calculate the intrapulmonary shunt before and after inhaled nitric oxide therapy. Intrapulmonary shunt was calculated from oxygen content (CO2) of different sites ( artery, mixed venous, alveolar capillary) by Fick equation:(CaO2-CcO2)/(CvO2-CcO2). A FiO2 of 1.0 and tidal volume of 6~8 ml/kg were chosen. Oxygen content was calculated from hemoglobin (Hb), oxygen saturation (SO2) and oxygen partial pressure (PO2) by the following equation: CO2 = 1.34*Hb*SO2 + 0,0031*PO2. PaO2, SaO2, PvO2 and SvO2 were measured from arterial and mixed venous blood samples taken from the radial arterial catheter and from the pulmonary artery catheter. ScO2 was estimated to be 1.0 with a FiO2 of 100%. PcO2 was considered to be the same as PAO2 (partial pressure of oxygen in the alveoli), and was calculated from the alveolar gas equation with PAO2 = [(atmospheric pressure - 47) * (FiO2)] - PaCO2/0.8.Other variables such as hemodynamic variables from pulmonary artery catheter were also collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Type A aortic dissection;
* After surgery;
* P/F ratio ≤ 200mmHg

Exclusion Criteria:

* Intracardiac shunt;
* Contradiction of PAC;
* Chronic pulmonary diseases before surgery;
* ECMO;
* Anticipation of death within 48 hours after operation;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: post-surgical type A aortic dissection patients with hypoxemia
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Intrapulmonary shunt with a PEEP of 5 cm H2O | 6 to 24 hours after surgery
  intrapulmonary shunt calculated by Fick equation with a PEEP of 5 cm H2O
Intrapulmonary shunt with a PEEP of 10 cm H2O | 30 minutes after increasing PEEP to 10cm H2O
  intrapulmonary shunt calculated by Fick equation with a PEEP of 10 cm H2O
Intrapulmonary shunt with a PEEP of 10 cm H2O and inhaled nitric oxide | 30 minutes after inhaling nitric oxide
  intrapulmonary shunt calculated by Fick equation with a PEEP of 10 cm H2O and inhaled nitric oxide
Intrapulmonary shunt with inhaled nitric oxide and a PEEP of 5 cm H2O | 30 minutes after decreasing PEEP to 5cm H2O
  intrapulmonary shunt calculated by Fick equation with inhaled nitric oxide and a PEEP of 5 cm H2O

SECONDARY OUTCOMES:
cardiac output collected from PAC with a PEEP of 5 cm H2O | 6 to 24 hours after surgery
  cardiac output in L/min
pulmonary artery pressure collected from PAC with a PEEP of 5 cm H2O | 6 to 24 hours after surgery
  pulmonary artery pressure in mmHg
pulmonary artery wedge pressure collected from PAC with a PEEP of 5 cm H2O | 6 to 24 hours after surgery
  pulmonary artery wedge pressure in mmHg
cardiac output collected from PAC with a PEEP of 10cm H2O | 30 minutes after increasing PEEP to 10cm H2O
  cardiac output in L/min
pulmonary artery pressure collected from PAC with a PEEP of 10 cm H2O | 30 minutes after increasing PEEP to 10cm H2O
  pulmonary artery pressure in mmHg
pulmonary artery wedge pressure collected from PAC with a PEEP of 10 cm H2O | 30 minutes after increasing PEEP to 10cm H2O
  pulmonary artery wedge pressure in mmHg
cardiac output collected from PAC with a PEEP of 10 cm H2O and inhaled nitric oxide | 30 minutes after inhaling nitric oxide
  cardiac output in L/min
pulmonary artery pressure collected from PAC with a PEEP of 10 cm H2O and inhaled nitric oxide | 30 minutes after inhaling nitric oxide
  pulmonary artery pressure in mmHg
pulmonary artery wedge pressure collected from PAC with a PEEP of 10 cm H2O and inhaled nitric oxide | 30 minutes after inhaling nitric oxide
  pulmonary artery wedge pressure in mmHg
cardiac output collected from PAC with inhaled nitric oxide and a PEEP of 5 cm H2O | 30 minutes after decreasing PEEP to 5 cm H2O
  cardiac output in L/min
pulmonary artery pressure collected from PAC with inhaled nitric oxide and a PEEP of 5 cm H2O | 30 minutes after decreasing PEEP to 5 cm H2O
  pulmonary artery pressure in mmHg
pulmonary artery wedge pressure collected from PAC with inhaled nitric oxide and a PEEP of 5 cm H2O | 30 minutes after decreasing PEEP to 5 cm H2O
  pulmonary artery wedge pressure in mmHg, etc

CONTACTS AND LOCATIONS:
Overall Officials: Guo-wei Tu, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hospital Fudan University, Shanghai, Shanghai Municipality, China